CLINICAL TRIAL: NCT03514472
Title: Impact of Dried Moringa Oleifera Leaves as Value Added Supplement in Enhancing Hemoglobin Status of Reproductive Aged Females of Low Socio-economic Group
Brief Title: Impact of Dried Moringa Oleifera Leaves in Enhancing Hemoglobin Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinnaird College for Women (Other)
Responsible Party: Principal Investigator, Madeeha Munir, Former Lecturer Minhaj University, Kinnaird College for Women
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MMunir
Record Dates: First submitted 2018-04-19; First posted 2018-05-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Anemia, Iron Deficiency
Keywords: Hb, Anemia,
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Intervention Model Description: In the study 34 of ages between 13-30 years divided into 2 age groups (below and above 18) were selected (excluding pregnant and lactating women) and were intervened with value added supplement " Moringa oleifera" for a period of three months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Below 18 years) (Active Comparator): Dried Moringa oleifera leaves (15g/recipe)
  Interventions: Dietary Supplement: Dried Moringa oleifera leaves
- Group B (Above 18) (Active Comparator): Dried Moringa oleifera leaves (15g/recipe)
  Interventions: Dietary Supplement: Dried Moringa oleifera leaves

INTERVENTIONS:
Dietary Supplement: Dried Moringa oleifera leaves

SUMMARY:
This research project is aimed at combating the nutritional deficiencies (Iron deficiency anemia) of reproductive aged females belonging to the underprivileged group of the society. Since anemia is one of the causes of still child-birth, preterm and low birth weight babies causing cognitive disabilities during the later years of life, So, it needs to be treated on priority bases.

DETAILED DESCRIPTION:
Mal-nutrition is a significant problem in the developing world, with serious consequences for human health and socio-economic development. It is estimated that over 43% women of reproductive age suffer from anemia. In Pakistan, about 35% non-pregnant and 51% pregnant women are suffering from anemia. Prevention and control against anemia rely on iron supplementation and food fortification on large scale. Both these methods are not affordable and feasible for poor people. Previous studies have shown that about 97% females do not meet their iron requirements. The possible reason to this can be iron losses from body including menstruation. To overcome these problems, culturally accepted, inexpensive and modified recipes were used to supply iron with addition of Moringa oleifera leaves (rich and cheap source of iron). In the study 34 of ages between 13-30 years were selected (excluding pregnant and lactating women) and were intervened with value added supplement " Moringa oleifera" for a period of three months. These recipes were made part of the diet by giving a dose of three meals per day on regular basis. Each recipe contained about 15 g of Dried Moringa powder. After the intervention, out of total 34, 3 females achieved normal Hb level of 12 g/dl. Overall, 94% cases of the study showed improvement of 1.8 g/dl (on average) in Hb level after intervention. There was a significant increase in blood Hb level (p<0.000) and both the var5iables were strongly and positively correlated (0.928). Variables of age and levels of education were weakly but significantly related to each other (p<0.001) in improving Hb after intervention.

Females with higher levels of education showed better response towards intervention.

After intervention with Moringa oleifera, an average increase of 1.5 g/dl in Hb was observed in the entire population whereas, members of Group B (ages above 18) showed more increase of 14.96% in their Hb level as compared to members of Group A (ages below 18) showing an increase of 12.96% in Hb level.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged females (13-30 years)

Exclusion Criteria:

* pregnant and Lactating women

Ages: 13 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Reproductive aged females ( those who are capable of bearing a child)
Enrollment: 34 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Improvement in Hemoglobin status | 3 months
  Comparison of Hb levels pre and post intervention

SECONDARY OUTCOMES:
Changes in BMI | 5 months
  Changes in BMI after improvement in Hb status

CONTACTS AND LOCATIONS:
Overall Officials: Madeeha Munir, M.Phil, Principal Investigator — Kinnaird College for Women

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anwar F, Bhanger MI. Analytical characterization of Moringa oleifera seed oil grown in temperate regions of Pakistan. J Agric Food Chem. 2003 Oct 22;51(22):6558-63. doi: 10.1021/jf0209894. PMID 14558778